CLINICAL TRIAL: NCT03423745
Title: Appropriate Number of Endotracheal Intubation Experience for First Attempt Successful Endotracheal Intubation During Cardiopulmonary Resuscitation
Brief Title: Appropriate Number of Endotracheal Intubation Experience for CPR
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Sang O, Park, Associate Professor, Konkuk University Medical Center
Other Study IDs: CPRintuexperience
Record Dates: First submitted 2017-12-25; First posted 2018-02-06 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Cardiopulmonary Arrest
Keywords: intubation; cardiopulmonary resuscitation; number of endotracheal intubation experience
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a clinical study based on analysis of video-clip data of intubation and clinical data for cardiopulmonary resuscitation patients between 2011.03.01.-2012.02.28.. Aim of this study is to estimate the appropriate number of endotracheal intubation(ETI) experience for successful ETI at first attempt during cardiopulmonary resuscitation.

DETAILED DESCRIPTION:
Endotracheal intubation(ETI) has been considered to be the best method of airway management during cardiopulmonary resuscitation(CPR). However, ETI during CPR requires high skill and experience. Therefore ETI during CPR should be performed by expert in ETI. But the definition of experts in ETI during CPR has not been done yet.

This study tried to estimate the appropriate number of ETI experience for successful ETI at first attempt during cardiopulmonary resuscitation. So the investigators analyze the success rate, speed, trial number, incidence of complications, and hands-off time of ETI using direct laryngoscopy (DL) which is standard device, in real clinical setting. In addition, this study analyze the residency training term, total number of ETI experience using DL at that time.

ELIGIBILITY:
Inclusion Criteria:

* patients who suffer sudden cardiac arrest

Exclusion Criteria:

* case of requesting the do-not-attempt resuscitation befor ETI
* intubated cases before arrival to emergency department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: emergency physicians in an urban ED at a tertiary training hospital in Seoul, Republic of Korea
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2012-02-29 (Actual); Study Completion 2012-02-29 (Actual)

PRIMARY OUTCOMES:
Successful intubation during CPR | successful endotracheal intubation with in 120 seconds
  endotracheal intubation, hands-off time < 10 seconds, first trial

CONTACTS AND LOCATIONS:
Overall Officials: Sang O Park, M.D., PhD, Principal Investigator — Department of Emergency Medicine, Konkuk University Medical center
Locations (1):
- Department of Emergency Medicine, Konkuk University Medical center, Seoul, South Korea

REFERENCES:
- [Background] Soar J, Nolan JP, Bottiger BW, Perkins GD, Lott C, Carli P, Pellis T, Sandroni C, Skrifvars MB, Smith GB, Sunde K, Deakin CD; Adult advanced life support section Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 3. Adult advanced life support. Resuscitation. 2015 Oct;95:100-47. doi: 10.1016/j.resuscitation.2015.07.016. No abstract available. PMID 26477701
- [Background] Wang HE, Simeone SJ, Weaver MD, Callaway CW. Interruptions in cardiopulmonary resuscitation from paramedic endotracheal intubation. Ann Emerg Med. 2009 Nov;54(5):645-652.e1. doi: 10.1016/j.annemergmed.2009.05.024. Epub 2009 Jul 2. PMID 19573949
- [Background] Je S, Cho Y, Choi HJ, Kang B, Lim T, Kang H. An application of the learning curve-cumulative summation test to evaluate training for endotracheal intubation in emergency medicine. Emerg Med J. 2015 Apr;32(4):291-4. doi: 10.1136/emermed-2013-202470. Epub 2013 Oct 23. PMID 24154942
- [Background] Mulcaster JT, Mills J, Hung OR, MacQuarrie K, Law JA, Pytka S, Imrie D, Field C. Laryngoscopic intubation: learning and performance. Anesthesiology. 2003 Jan;98(1):23-7. doi: 10.1097/00000542-200301000-00007. PMID 12502974